CLINICAL TRIAL: NCT05956951
Title: Restoring Spindle and Thalamocortical Efficiency in Early-Course Schizophrenia Patients Using Closed-Loop Auditory Stimulation
Brief Title: Restoring Spindle and Thalamocortical Efficiency in Early-Course Schizophrenia Patients Using Auditory Stimulation
Acronym: RESPITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fabio Ferrarelli (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Fabio Ferrarelli, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY20010236; R01MH130376 (NIH)
Record Dates: First submitted 2023-06-15; First posted 2023-07-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental: Night three- sham, night four - active (Experimental): This arm will receive sham auditory stimulation for the first 3 nights and active auditory stimulation for the fourth night.
  Night one - sham auditory stimulation, night 2 - sham auditory stimulation, night 3 - sham auditory stimulation, night 4 - active auditory stimulation
  Interventions: Device: Closed-loop auditory stimulation; Device: Sham auditory stimulation
- Experimental: Night three - active, night four - sham (Experimental): This arm will receive sham auditory stimulation for the first two nights, active auditory stimulation for the third night, and sham auditory stimulation for the fourth night.
  Night one - sham auditory stimulation, night two - sham auditory stimulation, night three - active auditory stimulation, night four - sham auditory stimulation
  Interventions: Device: Closed-loop auditory stimulation; Device: Sham auditory stimulation

INTERVENTIONS:
Device: Closed-loop auditory stimulation — Closed-loop auditory stimulation will be administered by a wearable EEG device (Philips SmartSleep Deep Sleep Headband). The EEG device will deliver auditory stimulation when slow-wave (deep) sleep is detected. Auditory stimulation will consist of 50ms long tones separated from each other by a fixed one-second inter-tone interval. The volume of each tone will be linearly modulated by sleep-depth such that louder (or softer) tones were played during deeper (or shallower) sleep.
Device: Sham auditory stimulation — Sham auditory stimulation consists of closed-loop auditory stimulation not being administered. A wearable EEG device (Philips SmartSleep Deep Sleep Headband) will not deliver closed-loop auditory stimulation and tones will not be played.

SUMMARY:
The purpose of this research is to identify differences in brain activity during sleep between health individuals and individuals with schizophrenia, schizophreniform, or schizoaffective disorder. This study will also investigate whether tones played during deep sleep can enhance specific features of sleep and whether enhancing such features is related to an improvement in cognitive performance.

DETAILED DESCRIPTION:
The overarching goal of the proposed study is to establish sleep spindle and slow wave abnormalities as early pathophysiological biomarkers of schizophrenia (SCZ). The investigators also seek to enhance spindle and slow wave deficits in EC-SCZ by utilizing a closed-loop auditory stimulation during sleep. The investigators will assess improvement of deficits with the use of a memory consolidation task before and after sleeping.

Participants will include early-course schizophrenia (EC-SCZ) subjects and healthy controls (HC). Participants will complete several assessments, including clinical evaluation, an IQ assessment (WASI), and at least 2 nights of sleep EEG recordings in the sleep clinic of UPMC Western Psychiatric Hospital with a polysomnography test (PSG) each night. Study participants will also fill out a Pittsburgh Sleep Quality Index (PSQI) which reports sleep habits. On one of the nights, EC-SCZ participants will receive active closed-loop auditory stimulation, while on another night they will receive sham closed-loop auditory stimulation. On all nights beside the adaptation night (night 1) participants will complete the motor sequence task (MST) and the AX-continuous performance task (AXCPT) before going to sleep. They will also repeat the task the following morning. There will be ~1 week between nights 2 and 3 and ~1 week between nights 3 and 4.

Aim 1. Establish sleep spindle and slow wave deficits in EC-SCZ patients relative to HC using a wireless ambulatory monitor.

H1a. EC-SCZ patients will have reduced sleep spindle duration and density compared to HC.

H1b. Slow wave density will be decreased in EC-SCZ patients relative to HC.

Aim 2. Determine that spindle and slow wave impairments can be acutely improved in EC-SCZ patients using closed-loop auditory stimulation during sleep.

H2a. Sleep spindle duration and density will increase during closed-loop auditory stimulation nights compared to baseline and sham intervention.

H2b. Slow wave density will increase during stimulation nights relative to baseline and sham intervention.

Aim 3. Examine the relationship between spindle and slow wave deficits and memory consolidation before and after their acute improvement in EC-SCZ patients relative to HC.

H3a. At baseline, sleep spindles and slow waves will predict memory consolidation in EC-SCZ patients and HC.

H3b. An increase in sleep spindles and slow waves during stimulating night will be associated with task-assessed memory consolidation improvement in EC-SCZ patients relative to baseline performance.

ELIGIBILITY:
Inclusion Criteria:

Early-course schizophrenia (EC-SCZ):

1. ages 18-40 years
2. current DSM-IV defined diagnosis of schizophrenia, schizophreniform or schizoaffective disorder, not drug-induced, with no previously reported psychotic episode
3. duration of ≤5 years from beginning of psychosis, defined by report of symptoms and/or history of treatment according to clinical guidelines employed in our University of Pittsburgh Medical Center (UPMC) psychoses clinics in Pittsburgh
4. lifetime exposure to antipsychotic medications ≤5 years

Healthy controls (HC):

1. ages 18-40 years
2. no lifetime history of psychiatric disorders
3. no first-degree family history of schizophrenia spectrum disorder or mood disorder with psychotic features.

Exclusion Criteria:

General exclusion criteria:

1. DSM-IV intellectual disability
2. significant head injury
3. medical illness affecting brain function or structure
4. pregnancy or postpartum (<6 weeks after delivery or miscarriage)
5. significant neurological disorder (e.g. seizure disorder)
6. inability to provide informed consent
7. current or past co-morbidity for alcohol or psychoactive substance dependence
8. substance abuse other than cannabis and/or alcohol within the past one year

For EC-SCZ:

a) a psychotic illness with a temporal relation to substance use or head injury

For healthy controls (HC):

1. difficult falling and/or staying asleep for more than half the nights of a week, on average
2. diagnosis of sleep apnea or restless leg syndrome
3. sleeping less than 5 hours or more than 10 hours daily, on average

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Deficits in sleep spindle and slow wave density in early-course schizophrenia patients (EC-SCZ). | baseline (pre closed-loop auditory stimulation)
  The difference between sleep spindle and slow wave density (measured as count per minute) in EC-SCZ relative to HC as recorded on a wireless ambulatory monitor.
Deficits in sleep spindle and slow wave duration in early-course schizophrenia patients (EC-SCZ). | baseline (pre closed-loop auditory stimulation)
  The difference between sleep spindle and slow wave duration (measured in seconds) in EC-SCZ relative to HC as recorded on a wireless ambulatory monitor.
Deficits in sleep spindle and slow wave amplitude in early-course schizophrenia patients (EC-SCZ). | baseline (pre closed-loop auditory stimulation)
  The difference between sleep spindle and slow wave amplitude (measured in microvolts) in EC-SCZ relative to HC as recorded on a wireless ambulatory monitor.
Improvement in sleep spindle and slow wave density. | baseline (pre closed-loop auditory stimulation), study completion (up to 6 weeks)
  Changes in sleep spindle and slow wave density (measured as count per minute) in EC-SCZ patients before and after closed-loop auditory stimulation during sleep.
Improvement in sleep spindle and slow wave duration. | baseline (pre closed-loop auditory stimulation), study completion (up to 6 weeks)
  Changes in sleep spindle and slow wave duration (measured in seconds) in EC-SCZ patients before and after closed-loop auditory stimulation during sleep.
Improvement in sleep spindle and slow wave amplitude. | baseline (pre closed-loop auditory stimulation), study completion (up to 6 weeks)
  Changes in sleep spindle and slow wave amplitude (measured in microvolts) in EC-SCZ patients before and after closed-loop auditory stimulation during sleep.
Relationship between spindle and slow wave deficits and memory consolidation. | baseline (pre closed-loop auditory stimulation), study completion (up to 6 weeks)
  Changes in task-assessed memory consolidation scores before and after closed-loop auditory stimulation in EC-SCZ compared to controls. Percent change in number of correct sequences in the morning compared to previous night on the Motor Sequence Tapping (MST) task will provide a proxy measure of overnight memory consolidation. Higher scores on the MST represent better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ferrarelli, MD,PhD, Principal Investigator — University of Pittsbrugh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with current National Institute of Mental Health (NIMH) data sharing rules as defined in NOT-MH-19-033 and will share all collected data in the National Database for Clinical Trials Related to Mental Illness (NDCT) database consistent with current guidelines and according to the schedule set in these guidelines.
Time Frame: Data will become available January 15th, 2024, and be updated every 6 months. Data will remain infinitely available.
Access Criteria: Everyone with a NIMH Data Archive login will be able to access the data.